CLINICAL TRIAL: NCT06622174
Title: Pulse Radiotherapy to Overcome Metastatic Immune System Evasion in Lung Cancer (PROMISE) - Phase I Trial
Brief Title: Pulse Radiotherapy to Overcome Metastatic Immune System Evasion in Lung Cancer
Acronym: PROMISE
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Houda Bahig (Other)
Collaborators: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor-Investigator, Houda Bahig, Radiation Oncologist, MD PhD, Centre hospitalier de l'Université de Montréal (CHUM)
Organization: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROMISE
Record Dates: First submitted 2024-09-21; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Non Small Cell Lung Cancer; Metastatic Lung Cancer
Keywords: Non small cell lung cancer; Metastatic lung cancer; Progressive disease; Polymetastatic; Immunotherapy resistance; Radiotherapy; Pulse radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulse Radiotherapy (Experimental): Pulsed radiotherapy combined with PD(L)-1 inhibitors targeting 2 to 5 progressive extracranial lesions per cycle
  Interventions: Radiation: Pulse radiotherapy

INTERVENTIONS:
Radiation: Pulse radiotherapy — Pulsed radiotherapy combined with PD(L)-1 inhibitors targeting 2 to 5 progressive extracranial lesions per cycle

SUMMARY:
This phase I study aims to evaluate the safety and effectiveness of adaptive pulsed radiotherapy combined with immunotherapy in patients with metastatic non-small cell lung cancer (NSCLC) resistant to immune checkpoint inhibitors. The primary goal is to assess treatment-related toxicity, while secondary objectives include progression-free survival, overall survival, and quality of life. The study will enroll 32 patients.

DETAILED DESCRIPTION:
Background: Non-small cell lung cancer (NSCLC) accounts for approximately 85% of all lung cancer cases and is a leading cause of cancer-related death globally. Despite the success of immune checkpoint inhibitors (ICIs) targeting PD-1 and PD-L1, many patients develop resistance to these therapies, either at the start (primary resistance) or over time (secondary resistance). This resistance leads to disease progression during or after treatment, posing a major clinical challenge. Recent studies suggest that combining ICIs with radiotherapy may improve treatment outcomes. Advances in pulsed radiotherapy, including stereotactic radiation cycles, have shown promising results in overcoming ICI resistance in metastatic disease.

Objective: This phase I prospective study aims to evaluate the safety (primary objective) and efficacy of pulsed radiotherapy in combination with PD(L)-1 inhibitors (with or without chemotherapy) in patients with polymetastatic NSCLC who have developed systemic resistance. The hypothesis is that this combination approach could improve patient outcomes by directly reducing tumor burden and enhancing the immune response, while maintaining an acceptable toxicity profile.

Methods: This single-arm phase I study will enroll 32 patients with NSCLC who show disease progression in ≥ 5 extracranial sites while on PD(L)-1 inhibitors (with or without chemotherapy). Pulsed radiotherapy will be delivered in up to 3 cycles, targeting 2 to 5 progressive lesions per cycle. Eligible participants must be 18 years or older, with systemic progression of NSCLC in ≥ 5 sites during treatment with ICIs, and an ECOG performance status of 0-2. Brain metastases are permitted but will not be included in the lesion count.

The primary endpoint is dose-limiting toxicity (DLT), defined by the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, focusing on grade 3-5 adverse events related to radiotherapy within 180 days of treatment. Secondary endpoints include the development of a clinical workflow for adaptive pulsed radiotherapy, progression-free survival (PFS), overall survival (OS), local recurrence, time to the next systemic treatment, and patient-reported quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 years old
* Ability to provide written informed consent
* Actively receiving PD(L)-1 inhibitors
* Progressive disease defined as per RECIST criteria 1.1 on CT metrics as a greater than 20% increase in the sum measurement of lesions, non-target unequivocal progressive disease or a new lesion on CT.
* Radiological progression to ≥ 5 disease sites. Progression at the primary tumor site should be counted within the total number of progressive lesions. For patients with lymph node metastases, each node is counted as one site of metastasis.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Patients with brain metastasis are allowed and should be treated as per standard of care
* All sites of disease can, in the opinion of the investigator, be safely treated and targetable with high-to-intermediate or low dose radiotherapy (taking into account prior local therapy, organ function and underlying medical condition such as inflammatory bowel disease, pulmonary fibrosis, etc.)
* Patients with prior metastases that have been treated with ablative therapies (e.g. radiotherapy, surgery or radiofrequency ablation) before their current line of systemic therapy, are eligible.
* Patients receiving additional systemic therapy agents such as chemotherapy are eligible, provided the other systemic agents are temporarily halted during radiation treatment.

Exclusion Criteria:

* Pregnant or breastfeeding individuals are excluded.
* Medical conditions that would hinder the safe administration of radiotherapy or follow-up.
* Patients who are ineligible for immunotherapy.
* Patients with a history of pneumonitis are excluded.
* Presence of an active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Toxicity | Within 180 days of radiotherapy completion
  Grade 3-5 toxicity as per Common Terminology Criteria for Adverse Events, version 4.0.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 years post radiotherapy
  Time from the start of adaptive pulse radiotherapy to the first documented disease progression or death from any cause.
Overall Survival (OS) | 2 years post radiotherapy
  Time from the start of treatment to death from any cause.
Quality of Life (QoL) | until 2 years after radiotherapy
  Measured using validated patient-reported outcome questionnaires, such as the EORTC QLQ-C30, at baseline, during treatment, and every 6 months.
Long term toxicity | More than 180 days post-treatment up to 2 year post treatment
  Grade 3-5 toxicity, based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided